CLINICAL TRIAL: NCT02200705
Title: Cryoablation of Low Risk Breast Cancer Less Than 1.5 cm: An Evaluation of Local Recurrence (Ice3 Trial)
Brief Title: Cryoablation of Low Risk Small Breast Cancer- ICE3 Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IceCure Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICMBC-02
Record Dates: First submitted 2014-07-22; First posted 2014-07-25 (Estimated); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: cryoablation, cryotherapy, breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- single arm, open label (Other): Early stage Breast cancers up to 1.5cm
  Interventions: Device: Ice-Sense3TM/ ProSenseTM

INTERVENTIONS:
Device: Ice-Sense3TM/ ProSenseTM

SUMMARY:
To evaluate the efficacy of cryoablation without lumpectomy and its impact on local and distant recurrence of early stage breast cancer .

ELIGIBILITY:
Inclusion Criteria:

1. Competent to sign informed consent
2. Diagnosis of invasive ductal breast carcinoma by core needle biopsy, meeting the following criteria:

   1. Unifocal primary disease NOTE: Patients with multifocal and/or multicentric in breast cancer, or evidence of EIC are NOT eligible. Patients with contralateral disease will remain eligible.
   2. Tumor size ≤1.5 cm in greatest diameter in the axis parallel to the treatment probe AND ≤1.5 cm in the axis anti-parallel to the treatment probe AND ≤1.5 cm in Anterior/ Posterior dimension. Tumor size ≤1.5 cm in greatest diameter as measured by breast ultrasound, mammogram and/or MRI. The largest dimension measured will be used to determine eligibility.
   3. Nottingham grade 1-2. Specifically, nuclear and mitotic scores must be less than or equal to 2.
   4. Estrogen receptor-positive, progesterone receptor-positive, HER2 negative
3. Age>= 50
4. Breast size adequate for safe cryoablation
5. Lesion must be sonographically visible at the time of treatment.
6. History of previously treated ipsilateral or contralateral breast carcinoma is not an exclusion criteria if the investigator is certain newly diagnosed carcinoma is new unifocal primary tumor.

Exclusion Criteria:

1. Presence of lobular carcinoma
2. Presence of luminal B pathology
3. Nottingham score of 3 (specially nuclear and mitotic score>2)
4. Presence of microinvasion, or invasive breast carcinoma with extensive intraductal component (EIC)
5. Presence of multifocal and/or multicentric in breast cancer
6. Presence of multifocal calcifications
7. Presence of prior or concurrent neoadjuvant chemotherapy for breast cancer
8. Presence of prior en bloc open surgical biopsy and/or lumpectomy for diagnosis/treatment of the index breast cancer
9. Patient that is not suitable to cryoablation procedure according to the physician opinion
10. ER AND PR negative, or Her2 positive noted on pre-cryo biopsy

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2024-03-17 (Actual); Study Completion 2024-05-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Ironwood Cancer & Research Centers, Glendale, Arizona
  - BreastLink, Santa Ana, California
  - Bridgeport Hospital, Yale Medical School, Trumbull, Connecticut
  - Dalton Surgical Group, Dalton, Georgia
  - Indiana University, Indianapolis, Indiana
  - Karmanos Cancer Institute, Detroit, Michigan
  - Regional Medical Imaging, Flint, Michigan
  - Comprehensive Breast Care, Troy, Michigan
  - CentraState Medical Center, Freehold, New Jersey
  - Breast Specialty care/ Presbyterian Hospital, Albuquerque, New Mexico
  - Mount Sinai Beth Israel, New York, New York
  - Columbia University/ NY Presbyterian hospital, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Montefiore Medical Center, New York, New York
  - Cincinnati Breast Surgeons Inc., Cincinnati, Ohio
  - University hospitals cleveland medical center, Cleveland, Ohio
  - Thomas Jefferson University hospital, Philadelphia, Pennsylvania
  - West Clinic, Germantown, Tennessee
  - Complete Breast Care, Plano, Texas

REFERENCES:
- [Derived] Jean J, Jochelson MS, Moo TA, Solomon SB, Bryce Y. Breast Cancer Recurrence after Cryoablation in Patients Who Are Poor Surgical Candidates or Who Refuse Surgery. J Vasc Interv Radiol. 2025 Jun;36(6):971-978. doi: 10.1016/j.jvir.2025.01.048. Epub 2025 Feb 3. PMID 39909175

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 19 sites in the USA. All study investigators had related experience in low-risk breast cancer treatment, imaging, and pathology assessments and were trained to perform the cryoablation procedure. The recruitment period lasted from October 2014 to February 2019.
Pre-assignment Details: A total of 212 Subjects were screened for enrollment in the study; 3 were screen failures, and 3 subjects withdrew consent before the procedure; 206 were enrolled and treated. Based on the DSMB recommendation, 12 subjects were excluded from the study after completing the cryoablation procedure. Nine (9) were due to deviation from inclusion criteria, and three (3) were due to incomplete treatment, resulting in the per-protocol study population of 194 subjects.
Groups:
- Single Arm, Open Label: Subjects with early-stage (up to 1.5 cm), low-risk breast cancer who met the eligibility criteria outlined in the study protocol were enrolled and underwent cryoablation using the IceCure Medical Ice-Sense3™/ProSense™ system.
Period: Overall Study
Arm/Group | Single Arm, Open Label
Started | 206
Per-protocol Study Population | 194
Completed | 131
Not Completed | 75
Not completed — Excluded | 12
Not completed — Death | 21
Not completed — Withdrawal by Subject | 22
Not completed — Lost to Follow-up | 13
Not completed — Physician Decision | 5
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: The primary analysis set includes 194 subjects (following the DSMB exclusion of 12 subjects).
Arm/Group | Single Arm, Open Label
Number analyzed (Participants) | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.9 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: African American | 14
  Ethnicity: Asian | 1
  Ethnicity: Caucasian | 160
  Ethnicity: Hispanic | 12
  Ethnicity: Native American | 2
  Ethnicity: Unknow | 5
Region of Enrollment [Number; unit: participants]
  United States | 194
Type of Tumor [Count of Participants; unit: Participants] — Subtype of breast cancer based on the cancer's molecular characteristics
  Participants
    Lumina A | 188
    Lumina B | 3
    Not specified | 3
ER (Estrogen Receptor) [Count of Participants; unit: Participants] — Lab assessment (IHC) of the percentage of estrogen receptors on breast cancer cells. ER-positive is defined when ≥1% of tumor cell nuclei stain positive.
  Participants
    Positive | 194
    Negative | 0
PR (Progesterone Receptor) [Count of Participants; unit: Participants] — Lab assessment (IHC) of the percentage of progesterone receptors on breast cancer cells. PR-positive is defined when ≥1% of tumor cell nuclei stain positive.
  Participants
    Positive | 180
    Negative | 14
Her2neu [Count of Participants; unit: Participants] — HER2 status is assessed by IHC to measure the amount of HER2 protein on the surface of breast cancer cells. HER2-negative is no staining or incomplete staining in >10% of cells. HER2-positive is strong complete staining in >10% of cells. HER2-negative breast cancer is a less aggressive form of cancer than HER2-positive cancers.
  Participants
    Positive | 0
    Negative | 194
Nottingham Grade (1-3) [Count of Participants; unit: Participants]
  Grade 1 (Low grade) - Least aggressive with good prognosis | 96
  Grade 2 (Intermediate-grade tumor) - Moderate aggressiveness and prognosis | 98

OUTCOME MEASURES:

1. Primary Outcome: Local Inbreast Breast Tumor Recurrence (IBTR) Rate
Description: 6 months post cryoabltion, then annually for 5 years
Time Frame: up to 5 years
Measure: Number (95% Confidence Interval); unit: Percentage of participants with IBTR
Arm/Group | Single Arm, Open Label
Number analyzed (Participants) | 194
Percentage of participants with IBTR | 4.3 [2.1 to 8.7]

2. Secondary Outcome: Complete Ablation of Primary Tumor
Description: Complete ablation of primary tumor up to 60 months after cryoablation
Time Frame: up to 5 years from procedure date.
Reporting Status: Not Posted

3. Secondary Outcome: Improvement or Maintenance of Subject's Quality of Life
Description: Quality of life will be assesed using NCCN DISTRESS THERMOMETER
Time Frame: at 6 months compare to the base line
Reporting Status: Not Posted

4. Secondary Outcome: Breast Cosmetics Satisfaction
Description: subjects and physician satisfaction from the cosmetic results
Time Frame: up to 5 years from procedure data.
Reporting Status: Not Posted

5. Secondary Outcome: Regional Recurrence Rate
Description: Regional Invasive breast tumor recurrence rate.
Time Frame: up to 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Distant Metastases Rate
Description: Distant metastases rate including contralateral Breast cancer
Time Frame: up to 5 years
Reporting Status: Not Posted

7. Secondary Outcome: Disease-free Survival (DFS)
Description: DFS from date of complete ablation of the primary tumor, until the first disease event where the disease event is defined as local (DCIS or invasive), regional, or distant breast cancer recurrence, second primary cancer, DCIS or invasive contralateral breast cancer, or death due to any cause
Time Frame: up to 5 years
Reporting Status: Not Posted

8. Secondary Outcome: Overall Survival
Description: Overall survival from the date of the cryoablation until the date of death from any cause or up to the 60 months follow up visit
Time Frame: up to 5 years
Reporting Status: Not Posted

9. Secondary Outcome: Breast Cancer Survival.
Description: Breast Cancer Survival from the date of cryoablation until the date of death from breast cancer or up to the 60 months follow-up visit.
Time Frame: up to 5 years
Reporting Status: Not Posted

10. Secondary Outcome: Adverse Events
Description: Adverse events related to study device or procedure rate
Time Frame: up to 2 years for AEs and up to 5 years for SAEs
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected through 2 years post-procedure, and serious adverse events (SAEs) were collected through the final follow-up (5 years post-procedure).
Arm/Group | Single Arm, Open Label
All-Cause Mortality (participants affected / at risk) | 21/206
Serious Adverse Events (participants affected / at risk) | 0/206
Other Adverse Events (participants affected / at risk) | 97/206
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm, Open Label (N=206)
Pain (General disorders) | 39 (41) — 39 events of local pain. 1 non-cardiac chest pain and 1 pain in extremity
Localized Edema (General disorders) | 39 (40)
Bruising (Injury, poisoning and procedural complications) | 61 (62)
Frost Injury (Injury, poisoning and procedural complications) | 5 (5) — Skin burn
Hematoma (Vascular disorders) | 9 (9)
Rash & Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Injection site reaction (General disorders) | 10 (11) — Including tenderness and skin reactions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT02200705/Prot_SAP_000.pdf